CLINICAL TRIAL: NCT02551926
Title: Health Education Using Text Messaging Prevents Hypertension in High Risk People: a Comparison Between Effectiveness of Electronic Text Messaging and Printed Material
Brief Title: Health Education Using Text Messaging Prevents Hypertension in High Risk People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, ِDirector of SDH center, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QUMS25
Record Dates: First submitted 2015-08-27; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (4):
- mobile text messaging (Experimental): Patients will receive some SMS in a regular interval.
  Interventions: Behavioral: mobile text messages; Device: mobile phone
- virtual communities (Experimental): Patients will receive some messages by a virtual community in a regular interval.
  Interventions: Behavioral: virtual community
- brochures (Experimental): Patients will receive some messages by as a printed media
  Interventions: Behavioral: brochures
- Control (Active Comparator): control group will be included without any intervention
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: mobile text messages
  Arms: mobile text messaging
Behavioral: virtual community
  Arms: virtual communities
Behavioral: brochures
  Arms: brochures
Other: Usual care
  Arms: Control
Device: mobile phone
  Arms: mobile text messaging

SUMMARY:
Prehypertension is a predisposing condition for morbidity inhypertension and cardiovascular diseases. Health education via electronic pathways such as mobile text messaging or virtual communities may provide more availability and adherence than printed media. Regarding lower costs of such electronic resources and continuity of interventions through these ways, assessing their effectiveness compared to a printed material may help health educators to choose proper methods for improve their educational attempts. Therefore, the current study aims to compare different tools for health education about healthy lifestyle in people with prehypertension. For this, educational interventions with similar content among 3 groups of people will be conducted (i.e., first group via mobile text messaging, second group using virtual communities, and third group by brochures as a printed media). A control group also will be considered without any intervention. Several phases are considered in the study. In phase 1 using health centers located in Qazvin city, people would be invited to a free screening program of prehypertension. Then, an eligible sample will be divided in three groups using a random allocation process (each one including 100-150 people with prehypertension). The blood pressure and health promotion lifestyle profile II (HPLP II) will be measured before intervention. A standard educational content using approaches of lifestyle promotion defined in HPLP II would be available for intervention groups during a time period of 1 month concurrently. At final phase, one month after termination of intervention blood pressure as primary outcome and lifestyle changes along with self-efficacy for lifestyle modification as secondary outcomes will be measured. This study may suggest effective ways for health education which is applicable by health care professionals to promote health status among peopleat risk of hypertension.

DETAILED DESCRIPTION:
Prehypertension is a predisposing condition for morbidity in hypertension and cardiovascular diseases. This has been defined as a systolic pressure from 120 to 139 mmHg or a diastolic pressure of 80-89 mm hg. The prevalence of this condition estimated to be at least 2 times higher than hypertension and those who have prehypertension 4 times more likely to progress to hypertension than normotensive people. Although, hypertension is a multi-factorial disease, lifestyle is associated mainly to its development. According to information, lifestyle changes may prevent more than 70% of primary hypertension and health education is a key strategy to promote lifestyle modification. Health education via electronic pathways such as mobile text messaging or virtual communities may provide more availability and adherence than printed media. Regarding lower costs of such electronic resources and continuity of interventions through these ways, assessing their effectiveness compared to a printed material may help health educators to choose proper methods for improve their educational attempts. Therefore, the current study aims to compare different tools for health education about healthy lifestyle in people with prehypertension. For this, educational interventions with similar content among 3 groups of people will be conducted (i.e., first group via mobile text messaging, second group using virtual communities, and third group by brochures as a printed media). A control group also will be considered without any intervention. Several phases are considered in the study. In phase 1 using health centers located in Qazvin city, people would be invited to a free screening program of prehypertension. Then, an eligible sample will be divided in three groups using a random allocation process (each one including 100-150 people with prehypertension). The blood pressure and health promotion lifestyle profile II (HPLP II) will be measured before intervention. A standard educational content using approaches of lifestyle promotion defined in HPLP II would be available for intervention groups during a time period of 1 month concurrently. At final phase, one month after termination of intervention blood pressure as primary outcome and lifestyle changes along with self-efficacy for lifestyle modification as secondary outcomes will be measured. This study may suggest effective ways for health education which is applicable by health care professionals to promote health status among people at risk of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* be >18 years
* have a diagnosis of prehypertension based on definition
* own a cell phone capable of receiving and sending text messages
* be a member of virtual communities
* Persian speaking
* willing to attend two data collection visits in Qazvin

Exclusion Criteria:

* admits to planning to terminate cell phone contract or excite form virtual communities during the next one month
* education less than primary school
* other major health problems (e.g., terminal stage of cancer, advanced liver disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Changes from baseline and 1 Months after the intervention

SECONDARY OUTCOMES:
changes in self-reported physical activity | Changes from baseline and 1 Months after the intervention
  Physical activity will be measured using a self-reported scale examining participants' self- reported physical activity for the past seven days. Six items
Changes in self-reported healthy eating | Changes from baseline and 1 Months after the intervention
  Healthy eating behavior will be measured using the Diet Guidelines Index (DGI). The DGI is a food-based dietary index that measures adherence to healthy eating recommendations over the previous month. It consists of 15 items that reflect current dietary guidelines,including consumption of vegetable and legumes, fruit, total cereals, meat, total dairy, beverages, sodium, saturated fat, alcoholic beverages, and added sugars. A diet quality score is obtained by summing the indicators of wholegrain cereals, lean meat, low-fat dairy, and dietary variety, and is informed by age- and sex-specific recommendations. Scores range from 0 to 150, with higher scores representing higher levels of healthy eating. Serving portions are described in the questionnaire, and participants were directed to refer to the healthy eating guidelines26 provided for further details.
Changes in self-reported Self-efficacy | Changes from baseline and 1 Months after the intervention
  Self-efficacy will be measured using the Medication Adherence Self-Efficacy Scale (MASES).he MASES is a patient-centered and self-administered questionnaire that consists of 26 items. The patient were asked to rate their confidence of taking antihypertensive medications in different conditions using a three-point scale

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - 22 Bahman Hospital, Qazvin, Qazvin Province
  - Qazvin University of Medical Sciences, Shahid Rajaei Hospital, Qazvin, Qazvin Province